CLINICAL TRIAL: NCT05747261
Title: An Open-Label, Non-Comparative Clinical Study of the Safety and Efficacy of an Adeno-Associated Viral Vector Carrying the SMN Gene (ANB-004 (JSC BIOCAD, Russia)) After a Single Intravenous Administration of Escalating Doses in Children With Spinal Muscular Atrophy
Brief Title: Study of the Safety and Efficacy of an Adeno-Associated Viral Vector Carrying the SMN Gene After a Single Intravenous Administration of Escalating Doses in Children With Spinal Muscular Atrophy (BLUEBELL)
Acronym: BLUEBELL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANB-004-1
Record Dates: First submitted 2023-02-14; First posted 2023-02-28 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Spinal Muscular Atrophy (SMA)
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: "3+3" design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Subjects in Cohort 1 will receive ANB-004 at a dose 1. Depending on the DLT, the cohort may include 1 to 6 subjects in the first stage and 9 to 12 in the second stage.
  Interventions: Genetic: ANB-004, dose 1
- Cohort 2 (Experimental): Subjects in Cohort 2 will receive ANB-004 at a dose 2. The dose for Cohort 2 will be determined at the IDMC meeting. Depending on the DLT, the cohort may include 1 to 6 subjects in the first stage and 9 to 12 in the second stage.
  Interventions: Genetic: ANB-004, dose 2
- Cohort 3 (Experimental): Subjects of Cohort 3, if included, will receive the drug at a dose 3. The dose for Cohort 3 will be determined at the IDMC meeting. Depending on the DLT, the cohort may include 1 to 6 subjects in the first stage and 9 to 12 in the second stage.
  Interventions: Genetic: ANB-004, dose 3

INTERVENTIONS:
Genetic: ANB-004, dose 1 — Adeno-associated viral vector carrying the SMN gene single infusion at dose 1. The duration of the infusion is about 60 minutes.
  Arms: Cohort 1
Genetic: ANB-004, dose 2 — Adeno-associated viral vector carrying the SMN gene single infusion at dose 2. The duration of the infusion is about 60 minutes.
  Arms: Cohort 2
Genetic: ANB-004, dose 3 — Adeno-associated viral vector carrying the SMN gene single infusion at dose 3. The duration of the infusion is about 60 minutes.
  Arms: Cohort 3

SUMMARY:
The goal of this multicenter, open-label, non-comparative, cohort study is to investigate the safety, immunogenicity, and efficacy of ANB-004 in children with spinal muscular atrophy. The study will have a standard 3+3 dose-escalation design.

DETAILED DESCRIPTION:
The study will be conducted in 2 stages:

Stage 1: pilot efficacy and safety study of different doses to select a potentially therapeutic dose for further study.

Stage 2: study of the efficacy and safety of ANB-004 at the selected potentially therapeutic dose.

At the first stage, the study will have a "3+3" design and involve dose escalation in two cohorts, with the possibility of including a third cohort. Three subjects are to be included in each cohort, each of whom will receive a pre-specified cohort dose of ANB-004 as a single intravenous infusion.

Subjects will be monitored for dose-limiting toxicity (DLT) events for 3 weeks after the drug infusion. In this study, DLT will include any of the CTCAE 5.0 grade 3 or higher adverse events (AEs) at least possibly related to the administration of the investigational product, except for an increase in body temperature at least possibly related to the administration of the investigational product, which will be classified as DLT starting from CTCAE 5.0 grade 4.

At the first stage, in the absence of DLT events in three subjects in the same cohort, an ID will be assigned, and an infusion will be administered to the first subject in subsequent cohort. If DLT events occur in 1 of 3 subjects in the same cohort, this cohort will additionally include 3 subjects who will receive the same ANB-004 dose with which the DLT event was observed. If DLT events occur in 2 or more of 3 subjects within the same cohort, the assignment of ID/infusion in subsequent subjects/study is suspended.

AT the second stage, if the IDMC judges that the potentially therapeutic dose was previously used in one of the cohorts, an additional 6 subjects will be included in this cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form for participation in the study signed by the subject's legal representative;
2. Subjects of either sex under the age of 240 days at the time of signing the Information Sheet for the Legal Representative of the Clinical Study Subject with Informed Consent Form;
3. A diagnosis of 5q-SMA (homozygous deletion of exon 7 of the SMN1 gene or heterozygous deletion of exon 7 + confirmed point mutation of the SMN1 gene) and 2 or 3 copies of the SMN2 gene established based on molecular genetic testing;
4. Subjects with 2 copies of the SMN2 gene can be included in the study both at the presymptomatic stage of the disease and in the presence of SMA symptoms. If symptoms are present, the age of onset of the disease should be up to 180 days from birth.
5. Subjects with 3 copies of the SMN2 gene can be included in the study if they have symptoms of SMA type 1 and the disease began before the age of 180 days.
6. The ability of the subject's legal representative, in the Investigator's opinion, to perceive information and follow the Protocol procedures

Exclusion Criteria:

1. A diagnosis of HIV infection, hepatitis B, hepatitis C, congenital syphilis in the study subject, as well as a documented diagnosis of HIV infection in the study subject's mother. Note: documented hepatitis B and/or hepatitis C and/or syphilis in the mother of a study subject is not an exclusion criterion in this clinical study, provided that standard breastfeeding rules are followed or the subject is not breastfed due to the low risk of transmission of hepatitis B and C viruses and Treponema pallidum from mother to child with breast milk;
2. Unwillingness of the legal representative to use alternative feeding methods (nasogastric tube, gastrostomy) in case of swallowing disorders and a risk of aspiration;
3. Anti-AAV9 antibody titer >1:50 determined by ELISA. Note: if a subject's screening anti-AAV9 antibody titer is >1:50, the anti-AAV9 antibody titer may be determined again. Subjects with anti-AAV9 antibody titers ≤1:50 in the second test may be included in the study;
4. Need for respiratory support for ≥16 hours per day or tracheostomy ;
5. Treatment with nusinersen, risdiplam, branaplam, onasemnogene abeparvovec or other antisense oligonucleotides/selective SMN2 splicing modifiers or gene therapy drugs for SMN1 transduction or other AAV-based gene therapy drugs regardless of serotype used previously (from birth) or planned for the main study period, i.e., within 12 months after the administration of the investigational product.
6. A need to use any medications for the treatment of myopathy or neuropathy, drugs for the treatment of diabetes, ongoing immunosuppressive therapy, or the need for immunosuppressive therapy after the start of the study (for example, glucocorticoids (except for premedication and post-medication), cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab, etc.);
7. Subjects with the following laboratory test results at screening:

   * increased activity of transaminases (ALT, AST) or GGT >2×ULN;
   * total bilirubin level ≥34 µmol/L;
   * creatinine level ≥160 µmol/L;
   * hemoglobin <80 g/L and >180 g/L;
   * WBC count >20x109/L;
   * Troponin I level > ULN.
8. Any concomitant diseases that, in the Investigator's opinion, may affect the safety of ANB-004 in the subject or have a significant impact on the assessment of the outcomes of SMA therapy;
9. A diagnosis of acute or chronic hepatic failure at screening;
10. A known allergy or intolerance to any components of the investigational product or pre- and post-medication drug (glucocorticoids);
11. Simultaneous participation of the subject in other clinical studies or previous participation in another clinical study using an experimental therapy.

Max Age: 240 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with adverse reactions | 12 months
Proportion of subjects with serious adverse reactions | 12 months
Proportion of subjects with CTCAE 5.0 or DAIDS grade 3 or higher adverse reactions | 12 months
  Since some of the severity criteria used in the CTCAE are not applicable to the pediatric population, it is proposed to use the 2017 Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events of the National Institute of Allergy and Infectious Diseases.
Time from date of birth to event | 12 months
  Time from date of birth to onset of a fatal event or the need for invasive respiratory support using tracheostomy or the need for non-invasive respiratory support for at least 16 hours a day for ≥14 consecutive days (in the absence of acute reversible disease and excluding surgery).
Motor development score | 12 months
  The assessment will be made using the motor development scale of a healthy child, which reflects the motor development milestones from birth to a certain age.
Change in the The Hammersmith Infant Neurological Examination (HINE) score | 12 months
  To assess the motor skills of study subjects, Section 2 of this scale will be used; the assessment will be made in subjects aged 3 to 24 months.

SECONDARY OUTCOMES:
Event occurrence | 12 months
  No fatal event, no need for invasive respiratory support using tracheostomy or non-invasive respiratory support for at least 16 hours a day for ≥14 consecutive days (in the absence of acute reversible disease and excluding surgery).
Documented evidence of efficacy | 12 months
  Changes in functional and motor abilities: percentage and age of children who can turn over and sit without support for more than 5, 10, 20 and 30 seconds on video records obtained during a visit to the study center and/or by a legal representative of the study participant outside the study center.

OTHER OUTCOMES:
Proportion of subjects with detectable IgM and IgG to the AAV9 protein capsid | 12 months
Proportion of subjects with detectable IgM and IgG to the SMN1 protein | 12 months
Proportion of subjects with detectable T cells specific to the AAV9 capsid | 12 months
Proportion of subjects with detectable T cells specific to the product of the SMN transgene | 12 months
Presence of the AAV9 vector in various body fluids (serum, saliva, urine, feces) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (6):
- 1. State Institution Republican Scientific and Practical Center "Mother and Child", Minsk, Belarus
- Russia (5):
  - Federal State Autonomous Educational Institution of Higher Education "N.I. Pirogov Russian National Research Medical University", Ministry of Health of the Russian Federation, Moscow
  - Federal State Autonomous Institution "National Medical Research Center for Children's Health", Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Educational Institution of Higher Education "St. Petersburg State Pediatric Medical University", Ministry of Health of the Russian Federation, Saint Petersburg
  - Federal State Budgetary Institution "V. A. Almazov National Medical Research Center" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - State Autonomous Healthcare Institution of the Sverdlovsk Region "Regional Children's Clinical Hospital", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No